CLINICAL TRIAL: NCT04295954
Title: Effect of a Semi-Presence Yoga Program, With Virtual Tutorized Home Tracking, on Dysmenorrhea in University Students: Randomized an Controlled Clinical Trial Protocol.
Brief Title: Effect of a Semi-Presence Yoga Program on Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Huelva (Other)
Responsible Party: Principal Investigator, Ana Abreu Sánchez, Teacher and Researcher, University of Huelva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DISMYOGA01
Record Dates: First submitted 2020-02-26; First posted 2020-03-05 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Dysmenorrhea Primary; Pain, Menstrual; Yoga
Keywords: clinical trial protocol; exercise therapy; quality of life; exercise movements technique; female
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Two groups will be formed with women who meet the inclusion criteria. Each participant will be randomly assigned to each group, receiving different treatment depending on the group in which it has been assigned: the intervention group will receive yoga intervention and the control group will continue with its conventional treatment for the dysmenorrhea.
Who Masked: Outcomes Assessor
Masking Description: The assignment to groups will be blind. A random number computer application will be awarded each participant to a group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Intervention (Experimental): This group will receive the Yoga Intervention for dysmenorrhea that will consist of 3 yoga sessions a week of 30 minutes each, for 12 weeks. The first 4 weeks 1 of the sessions will be face to face and the other 2 home sessions guided by a vieo and a brochure, and tutored from the virtual platform by the yoga teacher and researchers. This space will also serve for participants to share experiences.
  After the first 4 weeks, participants will continue with the virtually tutored home yoga program, consisting of 3 weekly sessions of 30 minutes until completing the 12 weeks. They will be protected in all cases by the teacher and researchers.
  All intervention group participants will be invited to participate in online focus groups during week 12 to explore their experiences and satisfaction with the progress of the study and to implement adaptations, if necessary.
  They will be evaluated before the start of the yoga program per month, 3 months, 6 months and a year after the intervention.
  Interventions: Other: Yoga Intervention
- Control group without intervention (No Intervention): Participants in the comparison group without intervention will not receive yoga intervention, will follow their conventional treatment and their usual daily activities. They will be told not to do yoga. They will be evaluated in advance, per a month, 3 months, 6 months and a year after the intervention.

INTERVENTIONS:
Other: Yoga Intervention — It is an intervention based on Hatha yoga designed specifically to improve dysmenorrhea. This intervention consists of physical postures, also called asanas; meditation and breathing. It begins with a progression of various asanas until reaching the three central postures: "cat, cobra and fish". The compensation asanas of these central postures are then performed, and it is closed with a relaxation. The program and Yoga Intervention have been triangulated by experts and piloted afterwards.
  Arms: Yoga Intervention

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a blended learning yoga program using virtually tutored home follow-up on pain intensity measured using the VAS scale, quality of life and adherence among nursing students with moderate to severe dysmenorrhea, compared to a control group of students.

Half of the women involved will receive a yoga intervention for dysmenorrhea for 12 weeks, while the other half will continue with their conventional treatment during the same period. The results of the evaluations carried out prior, to the month, 3 months, 6 and 12 months of the intervention will be compared.

DETAILED DESCRIPTION:
Dysmenorrhea affects between 50% and 90% of women of childbearing age worldwide, the figure is estimated to be 74.8% in Spain. In addition to pain, other menstrual symptoms affect the normality of those with it, and it is found to cause absenteeism at work and school and influence academic performance. Self-medication with painkillers is one of the most used self-care measures by women with dysmenorrhea despite not being the most appropriate. So, in recent decades new lines are being investigated that can help reduce the impact of the problem on women with dysmenorrhea.

According to several studies, physical exercise is an effective supportive therapy in dysmenorrhea, and in particular through yoga has been found relief from menstrual symptoms and associated anguish, and improvement in pain and quality of life. The practice of yoga has shown physical, emotional and general well-being improvements. But it is advisable to continue to investigate because of the heterogeneity if the interventions it is difficult to reach consensus as to the time and frequency of the sessions, program duration or type of yoga program and the most appropriate postures. It is therefore recommended to unify the characteristics of the participants, describe the programs in detail, extend the duration of clinical trials, and carry them out with greater methodological rigor.

A novel aspect of this specific yoga program for dysmenorrhea is the semi-presence and home virtual tutoring of the intervention that will make it easier for women to practice at home according to their time possibilities or their health status, being guided by experts and supported with validated material for the intervention. Online tutoring and monitoring can promote adherence, compliance with intervention more rigorously, and even use of more advisable self-care measures, as evidenced by previous studies with patients with other health problems.

So, the aim of this clinical trial is to analyze the effects of a 12-month Hatha Yoga program based on physical postures, breathing and meditation in a blended learning modality with a virtually tutored home follow-up, on the intensity of pain measured using the VAS and on the quality of life of nursing students with dysmenorrhea in Andalusia. The results will be compared with a control group of students who will continue their usual lifestyle during the same period. They will be evaluated in advance, within a month, 3 months, 6 months and one year after receiving the intervention. The project has been approved by the Andalusian Ethics and Research Committee.

The yoga program has been designed according to previous studies for dysmenorrhea and the Guidelines for Developing Yoga Interventions for Randomized Trials. It is a Hatha Yoga Intervention for dysmenorrhea, i.e. body, respiratory and mental work led by teachers with more than 600 hours of accredited training and at least 300 hours of experience with adults with varied chronic health conditions. The program has been triangulated by experts and piloted after. It will be held at the Centre of Physical and Sports Activities of the El Carmen University Campus of the University of Huelva. The intervention consists of three weekly 30-minute yoga sessions for 12 weeks. The first 4 weeks 1 face to face session and 2 home yoga sessions guided by the yoga teacher will be taught weekly in all cases. At home, the participants will also have a video and a diptych of the same yoga series designed for this trial. There will be a virtual platform to project participants by the yoga teacher and researchers. After the first 4 weeks they will continue with 3 weekly sessions of 30 minutes each, of directed home yoga also. All intervention group participants will be invited to participate in online focus groups during week 12 of the clinical trial to explore their experiences and satisfaction with the progress of the study and to implement adaptations, if necessary. Each session consists of physical postures or preparation asanas, and they are a means to reach the central asanas "cobra, cat and fish". Followed by asanas of compensation, relaxation and meditation.

Our hypothesis is that women who participate in a blended Hatha Yoga program will report an improvement in their intensity of pain and the symptoms associated with dysmenorrhea, quality of life, absenteeism, academic performance, daytime fatigue, stress, wellbeing, among other secondary results in the short, mid and long term

ELIGIBILITY:
Inclusion Criteria:

• Nulliparous women who exhibit moderate-severe pain, 4-10 according to VAS, associated with menstruation in their last cycle, have no history of diagnosed gynecological pathology, and have an internet access device (mobile, computer or table).

Exclusion Criteria:

• Those who do not meet the criteria for inclusion or do not wish to participated voluntarily, suffer from any other illnesses associated with pain or limiting physical exercise, as well as exclude women who already perform yoga.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female, nulliparous
Enrollment: 50 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain Intensity | Change from baseline pain intensity at 1 month; Change from baseline pain intensity at 3 months; Change from baseline pain intensity at 6 months; Change from baseline pain intensity at 12 months;
  Pain intensity will be assessed with the Visual Analog Pain Scale (VAS): Is a continuous scale consisting of a horizontal line of 10 centimeters (100 mm) in length, ranging "painless" (score of 0) to "pain as severe as it could be" or "worst imaginable pain" (score of 100).
Changes in Satisfaction and Quality of life | Change from baseline Quality of Life at 1 month; Changes from baseline Quality of Life at 3 months; Changes from baseline Quality of Life at 6 months; Changes from baseline Quality of Life at 12 months.
  Quality of life will be evaluated with the SF-12 Abbreviated Quality of Life Questionnaire, with consists of 12 quality of life items measured o a Likert scale between 0 and 6. Explore multidimensional health and self-administer.

SECONDARY OUTCOMES:
Sleep quality | baseline,1 month, 3 months, 6 months, 12 months
  Sleep quality will be measured with the Pittsburgh Sleep Quality Index (PSQI). It is a self-report scale that is completed in 5 minutes; it consists of 19 items and contains seven subscales each weighted equally on a scale of 0 to 3, with higher scores indicating a lower sleep quality rating. The total sum ranging from 0 (good sleep quality) to 21 (poor sleep quality) reflects poor sleep if it is ≥ 5.
Degree of drowsiness | baseline, 1 month, 3 months, 6 months, 12 months
  Degree of drowsiness will be measured with the Epworth Sleepiness Questionnaire (ESE), a self-applicable instrument for assessing the propensity to fall asleep in eight situations. Each is evaluated on a scale of 0-3, where 0 means zero probability of falling asleep and 3 high probability. The sum of the grades results: 0-24.
Anxiety State | baseline, 1 month, 3 months, 6 months, 12 months
  Anxiety as a state, will be measured using the STAI Status Scale, Spielberger. Will assesse how an individual feels at a given time. The scale include 20 items using a 4-points Likert scale (20 to 80). Higher scores indicate an increase in anxiety levels.
Anxiety Traits | baseline, 1 month, 3 months, 6 months, 12 months
  Anxiety as a trait, will be measured using the STAI Spielberger Trait. Anxiety traits will assesse how an individual feels in general. Include 20 items using a 4-points Likert scale (20 to 80). Higher scores indicate an increase in anxiety levels.
Stress | baseline, 1 month, 3 months, 6 months, 12 months
  Stress will be measured with the Perceived Stress Scale (PSS), is a self-reporting instrument that assesses the perceived stress level over the last month, consists of 14 items ith a five points scale response format (0= never, 1= almost never, 2= from time to time, 3= often, 4= very often). The highest score corresponds to a higher level of perceived stress.
Degree of change | baseline, 1 month, 3 months, 6 months, 12 months
  The perception of degree of change on the overall state will be measured with the Grade of Change Perception Scale (GAC), with the following gradation "Much worse/ worse /a little better / same / a little better/ better" until "much better".
Perceived well-being | baseline, 1 month, 3 months, 6 months, 12 months
  Well-being will be measured by the Spanish version of the Warwick-Edinburgh Mental Welfare Scale (EBMWE). The questionnaire has 14 items, with 5 answer options (from 1 to 5). Higher scores indicate better mental well-being.
Menstrual symptoms | baseline, 1 month, 3 months, 6 months, 12 months
  It will be evaluated with 13 closed dichotomous questions, about presence or absence of vomiting, dizziness, headaches, irritability, edema, headaches, constipation, diarrhea, tiredness, anxiety among others.
Menstrual Attitude | baseline, 1 month, 3 months, 6 months, 12 months
  It will be evaluated using the MAQ (Brooks-Gunn & Ruble 1980) Menstrual Attitude Questionnaire. The Mentrual Attitude Questionnaire is a useful tool for evaluating menstrual attitudes among high school and college students. It consists of 7 answer options, in which 1 means "totally disagree" and 7 "totally agree". It is self-administered.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Abreu Sánchez, PhD, Study Director — Universidad de Huelva, Facultad de Enfermería
Locations (1):
- Ana Abreu Sánchez, Huelva, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iacovides S, Avidon I, Baker FC. What we know about primary dysmenorrhea today: a critical review. Hum Reprod Update. 2015 Nov-Dec;21(6):762-78. doi: 10.1093/humupd/dmv039. Epub 2015 Sep 7. PMID 26346058
- [Background] Fernandez-Martinez E, Onieva-Zafra MD, Parra-Fernandez ML. Lifestyle and prevalence of dysmenorrhea among Spanish female university students. PLoS One. 2018 Aug 10;13(8):e0201894. doi: 10.1371/journal.pone.0201894. eCollection 2018. PMID 30096156
- [Background] McGovern CE, Cheung C. Yoga and Quality of Life in Women with Primary Dysmenorrhea: A Systematic Review. J Midwifery Womens Health. 2018 Jul;63(4):470-482. doi: 10.1111/jmwh.12729. Epub 2018 Jun 14. PMID 29902363
- [Background] Fernandez-Martinez E, Onieva-Zafra MD, Parra-Fernandez ML. The Impact of Dysmenorrhea on Quality of Life Among Spanish Female University Students. Int J Environ Res Public Health. 2019 Feb 27;16(5):713. doi: 10.3390/ijerph16050713. PMID 30818861
- [Background] Armour M, Smith CA, Steel KA, Macmillan F. The effectiveness of self-care and lifestyle interventions in primary dysmenorrhea: a systematic review and meta-analysis. BMC Complement Altern Med. 2019 Jan 17;19(1):22. doi: 10.1186/s12906-019-2433-8. PMID 30654775
- [Background] Armour M, Ee CC, Naidoo D, Ayati Z, Chalmers KJ, Steel KA, de Manincor MJ, Delshad E. Exercise for dysmenorrhoea. Cochrane Database Syst Rev. 2019 Sep 20;9(9):CD004142. doi: 10.1002/14651858.CD004142.pub4. PMID 31538328
- [Background] Ross A, Thomas S. The health benefits of yoga and exercise: a review of comparison studies. J Altern Complement Med. 2010 Jan;16(1):3-12. doi: 10.1089/acm.2009.0044. PMID 20105062
- [Background] Cramer H, Lauche R, Anheyer D, Pilkington K, de Manincor M, Dobos G, Ward L. Yoga for anxiety: A systematic review and meta-analysis of randomized controlled trials. Depress Anxiety. 2018 Sep;35(9):830-843. doi: 10.1002/da.22762. Epub 2018 Apr 26. PMID 29697885
- [Background] McCall MC, Ward A, Roberts NW, Heneghan C. Overview of systematic reviews: yoga as a therapeutic intervention for adults with acute and chronic health conditions. Evid Based Complement Alternat Med. 2013;2013:945895. doi: 10.1155/2013/945895. Epub 2013 May 16. PMID 23762174
- [Background] Dodich A, Zollo M, Crespi C, Cappa SF, Laureiro Martinez D, Falini A, Canessa N. Short-term Sahaja Yoga meditation training modulates brain structure and spontaneous activity in the executive control network. Brain Behav. 2019 Jan;9(1):e01159. doi: 10.1002/brb3.1159. Epub 2018 Nov 28. PMID 30485713
- [Background] Kim SD. Yoga for menstrual pain in primary dysmenorrhea: A meta-analysis of randomized controlled trials. Complement Ther Clin Pract. 2019 Aug;36:94-99. doi: 10.1016/j.ctcp.2019.06.006. Epub 2019 Jun 25. PMID 31383452
- [Background] Yonglitthipagon P, Muansiangsai S, Wongkhumngern W, Donpunha W, Chanavirut R, Siritaratiwat W, Mato L, Eungpinichpong W, Janyacharoen T. Effect of yoga on the menstrual pain, physical fitness, and quality of life of young women with primary dysmenorrhea. J Bodyw Mov Ther. 2017 Oct;21(4):840-846. doi: 10.1016/j.jbmt.2017.01.014. Epub 2017 Feb 7. PMID 29037637
- [Background] Armour M, Parry K, Al-Dabbas MA, Curry C, Holmes K, MacMillan F, Ferfolja T, Smith CA. Self-care strategies and sources of knowledge on menstruation in 12,526 young women with dysmenorrhea: A systematic review and meta-analysis. PLoS One. 2019 Jul 24;14(7):e0220103. doi: 10.1371/journal.pone.0220103. eCollection 2019. PMID 31339951
- [Background] Collins SL, Moore RA, McQuay HJ. The visual analogue pain intensity scale: what is moderate pain in millimetres? Pain. 1997 Aug;72(1-2):95-7. doi: 10.1016/s0304-3959(97)00005-5. PMID 9272792
- [Background] Sherman KJ. Guidelines for developing yoga interventions for randomized trials. Evid Based Complement Alternat Med. 2012;2012:143271. doi: 10.1155/2012/143271. Epub 2012 Oct 2. PMID 23082079
- [Background] Jeter PE, Slutsky J, Singh N, Khalsa SB. Yoga as a Therapeutic Intervention: A Bibliometric Analysis of Published Research Studies from 1967 to 2013. J Altern Complement Med. 2015 Oct;21(10):586-92. doi: 10.1089/acm.2015.0057. Epub 2015 Jul 21. PMID 26196166
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Ferrer M, Vilagut G, Monasterio C, Montserrat JM, Mayos M, Alonso J. [Measurement of the perceived impact of sleep problems: the Spanish version of the functional outcomes sleep questionnaire and the Epworth sleepiness scale]. Med Clin (Barc). 1999 Sep 11;113(7):250-5. Spanish. PMID 10544379
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Lopez MA, Gabilondo A, Codony M, Garcia-Forero C, Vilagut G, Castellvi P, Ferrer M, Alonso J. Adaptation into Spanish of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) and preliminary validation in a student sample. Qual Life Res. 2013 Jun;22(5):1099-104. doi: 10.1007/s11136-012-0238-z. Epub 2012 Jul 27. PMID 22836376
- [Background] Castellvi P, Forero CG, Codony M, Vilagut G, Brugulat P, Medina A, Gabilondo A, Mompart A, Colom J, Tresserras R, Ferrer M, Stewart-Brown S, Alonso J. The Spanish version of the Warwick-Edinburgh mental well-being scale (WEMWBS) is valid for use in the general population. Qual Life Res. 2014 Apr;23(3):857-68. doi: 10.1007/s11136-013-0513-7. Epub 2013 Sep 5. PMID 24005886
- [Result] Cramer H, Ward L, Saper R, Fishbein D, Dobos G, Lauche R. The Safety of Yoga: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Am J Epidemiol. 2015 Aug 15;182(4):281-93. doi: 10.1093/aje/kwv071. Epub 2015 Jun 26. PMID 26116216
- [Result] Matthewman G, Lee A, Kaur JG, Daley AJ. Physical activity for primary dysmenorrhea: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2018 Sep;219(3):255.e1-255.e20. doi: 10.1016/j.ajog.2018.04.001. Epub 2018 Apr 7. PMID 29630882